CLINICAL TRIAL: NCT06429800
Title: A Phase 1 Study to Evaluate the Safety and Preliminary Efficacy of ATA3219, Allogeneic Anti-CD19 Chimeric Antigen Receptor T-cell (CAR T) Therapy, in Subjects With Systemic Lupus Erythematosus
Brief Title: A Study to Evaluate the Safety and Preliminary Efficacy of ATA3219 in Participants With Systemic Lupus Erythematosus
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Financial
Sponsor: Atara Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ATA3219-AEC-104
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Lupus Nephritis; Systemic Lupus Erythematosus
Keywords: Lupus Nephritis (LN); Systemic Lupus Erythematosus (SLE); Anti CD19 Chimeric Antigen Receptor T cell (CAR T) Therapy; Human leukocyte antigen (HLA); Epstein-Barr virus (EBV) T cells; Extrarenal Systemic Lupus Erythematosus (ERL)
MeSH Terms: conditions — Lupus Nephritis; Lupus Erythematosus, Systemic; Epstein-Barr Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Cohort LN: ATA3219 Dose Level -1 (Experimental): Participants will receive a single IV infusion of ATA3219 Dose Level -1 (if required) on Day 1 of a 28-day dose limiting toxicity (DLT) observation period.
  Interventions: Drug: ATA3219
- Cohort LN: ATA3219 Dose Level 1 (Experimental): Participants will receive a single IV infusion of ATA3219 Dose Level 1 on Day 1 of a 28-day DLT observation period.
  Interventions: Drug: ATA3219
- Cohort LN: ATA3219 Dose Level 2 (Experimental): Participants will receive a single IV infusion of ATA3219 Dose Level 2 on Day 1 of a 28-day DLT observation period.
  Interventions: Drug: ATA3219
- Cohort LN: ATA3219 Dose Level 3 (Experimental): Participants will receive a single IV infusion of ATA3219 Dose Level 3 on Day 1 of a 28-day DLT observation period.
  Interventions: Drug: ATA3219
- Cohort ERL: ATA3219 Dose Level -1 (Experimental): Participants will receive a single IV infusion of ATA3219 Dose Level -1 (if required) on Day 1 of a 28-day DLT observation period.
  Interventions: Drug: ATA3219
- Cohort ERL: ATA3219 Dose Level 1 (Experimental): Participants will receive a single IV infusion of ATA3219 Dose Level 1 on Day 1 of a 28-day DLT observation period.
  Interventions: Drug: ATA3219
- Cohort ERL: ATA3219 Dose Level 2 (Experimental): Participants will receive a single IV infusion of ATA3219 Dose Level 2 on Day 1 of a 28-day DLT observation period.
  Interventions: Drug: ATA3219
- Cohort ERL: ATA3219 Dose Level 3 (Experimental): Participants will receive a single IV infusion of ATA3219 Dose Level 3 on Day 1 of a 28-day DLT observation period.
  Interventions: Drug: ATA3219

INTERVENTIONS:
Drug: ATA3219 — ATA3219 is an allogeneic chimeric antigen receptor (CAR) T-cell therapy containing a second generation CD19 CAR construct in Epstein Barr virus (EBV) T cells, administered intravenously on Day 1.

SUMMARY:
The purpose of the study is to evaluate the safety and preliminary efficacy of ATA3219 for treatment of participants with lupus nephritis (LN) following lymphodepletion (LD) and in participants with extrarenal systemic lupus erythematosus (SLE) without LD.

DETAILED DESCRIPTION:
This is a Phase 1, multi-centered, open-labeled, dose escalation study to evaluate the safety and preliminary efficacy of ATA3219 (as monotherapy) in participants with LN following LD (Cohort LN) and in participants with extrarenal SLE (ERL) without LD (Cohort ERL). This study is planned to be conducted in the United States, Canada, and Australia. For each cohort, up to 3 dose levels (DLs) will be explored in the dose escalation portion of the study and if needed a lower dose may be explored. Prior to undergoing any screening procedure, prospective participants must undergo the ATA3219 inventory check assessments to ensure availability of an appropriate partially human leukocyte antigen (HLA)-matched ATA3219 product lot. Before administration of ATA3219, participants will receive LD treatment (Cohort LN) or methylprednisolone treatment (Cohort ERL). For all enrolled participants, hospitalization during and following ATA3219 dosing is mandatory. Participants will receive a single dose intravenous (IV) infusion of ATA3219 (monotherapy) on Day 1. Participants will remain inpatient for a minimum of 1 week post ATA3219 dosing, where they will be frequently monitored. Clinical responses will be assessed by the investigator on Day 28 (+ 5 days) following each dose of ATA3219. For each cohort, during dose escalation, up to 3 DLs of ATA3219 are planned to be evaluated sequentially and a lower dose may be added. At least 3 and up to 6 dose-limiting toxicity (DLT)-evaluable participants, those who complete the 28-day DLT observation period, will be assessed at each DL. Within each DL, treatment will be staggered to allow appropriate safety monitoring by an independent Data Safety Monitoring Committee (DSMC).

Enrolled participants who do not receive ATA3219 for any cause (e.g., rapid deterioration) will be replaced. Participants who experience an adverse event (AE) during the 28-day DLT observation and complete the observation period will not be replaced. In addition, if a participant is treated with ATA3219 and discontinues for any reason other than due to a DLT prior to completing the 28-day DLT observation period, an additional participant may be enrolled at the dose level to ensure that the recommended phase 2 dose (RP2D) can be determined, with a goal not to exceed 6 participants treated/dose level. In rare situations, retreatment of participants with inadequate renal response may be considered.

After treatment is completed or discontinued, participants will be followed for safety and clinical response for up to 24 months from the last dose of ATA3219. A separate long-term follow-up study will be conducted to follow participants for up to a total of 15 years after their last dose of ATA3219.

ELIGIBILITY:
Inclusion Criteria for all Participants:

1. Diagnosed with SLE according to the 2019 European League Against Rheumatism/American College of Rheumatology classification for SLE OR the Systemic Lupus International Collaborating Clinics Classification criteria [Petri 2012].
2. Meets one or more of the following immunologic criteria during screening:

   1. Anti double stranded DNA above laboratory reference range, except enzyme linked immunosorbent assay (2 × above laboratory reference range), OR
   2. Presence of one or more of following autoantibodies: anti-Smith, anti-ribonucleoprotein, or anti-phospholipid, OR
   3. Low complement as demonstrated by low complement component 3, low complement component 4, or low complement CH50.
3. Adequate lung, liver, kidney, and cardiac function.

   Inclusion Criteria for Cohort LN Only:
4. History of International Society of Nephrology (ISN)/Renal Pathology Society (RPS) Class III or IV with or without Class V glomerulonephritis on renal biopsy either within 6 months prior to screening or as performed during screening. Biopsy should demonstrate evidence of active nephritis.
5. Proteinuria level between ≥ 1.0 to 6.0 g/g via urine protein creatinine ratio during screening.
6. Has refractory LN defined as having received 1 or more standard therapies for LN (which must have included mycophenolate mofetil, mycophenolic acid, or cyclophosphamide), and:

   1. Has worsening LN (per criteria listed in [Gordon 2009]) while on treatment, OR
   2. Has not achieved a complete renal response (CRR) after 2 or more lines of therapy, OR
   3. Has not achieved a CRR after first-line therapy after a minimum of 12 months.

   Inclusion Criteria for Cohort Extrarenal SLE Only:
7. Hybrid SELENA-SLEDAI score of ≥ 8 points at screening

   * For participants with BILAG A involvement, this must include "clinical" hybrid SELENA-SLEDAI score of ≥ 4 points
   * For participants without BILAG A involvement, this must include clinical hybrid SELENA-SLEDAI score of ≥ 6 points
8. Meets BILAG-2004 criteria: At least 1 of the following:

   * BILAG-2004 level A disease in ≥ 1 organ system
   * BILAG-2004 level B disease in ≥ 2 organ systems and physician global assessment score ≥ 2
9. Persistent disease activity as defined in inclusion criterion #8 (above), despite having received 2 or more standard-of-care immunosuppressive therapies for SLE (as determined by the investigator), which may include biologics, for a minimum of 3 months (for participants with BILAG A involvement in any organ systems) or a minimum of 6 months (for participants with only BILAG B involvement in ≥ 2 organ systems).

Exclusion Criteria for all Participants:

1. Has a concurrent systemic autoimmune disease that may confound study assessments other than SLE, LN, or cutaneous lupus erythematosus.
2. Has any unstable or progressive manifestation of SLE that is likely to warrant an intensification of lupus-directed therapy
3. Has a history of catastrophic antiphospholipid syndrome, or any history of prior thrombosis due to antiphospholipid syndrome resulting in hospitalization due to myocardial infarction, pulmonary embolism, or stroke.
4. Has a history of bleeding disorder requiring hospitalization or systemic therapeutic intervention within the previous 3 months, or for participants without a prior kidney biopsy meeting eligibility criterion within the past 6 months who will require a biopsy during screening, any contraindication to kidney biopsy.
5. Presence of clinically relevant (as assessed by the investigator) central nervous system (CNS) pathology such as epilepsy, seizure, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis; any BILAG A CNS manifestation within 4 weeks of enrollment.
6. Any prior cellular therapies, obinutuzumab, anti-cluster of differentiation 19 (CD19) antibody, or B-cell targeting bispecific antibody, unless B-cells have recovered to baseline as assessed by the investigator. Investigational therapies or initiation of new SLE-directed therapies within 4 weeks.

   Exclusion Criteria for Cohort LN Only:
7. Severe kidney disease as assessed locally, defined as history of ISN/RPS Class VI or isolated Class V glomerulonephritis (without co existent/predominant Class III or IV glomerulonephritis) on renal biopsy.
8. Known hypersensitivity to fludarabine or cyclophosphamide.
9. Any inability to discontinue or taper systemic SLE therapy prior to infusion of ATA3219, including

   1. Tapering of corticosteroids to ≤ 10 mg/day and
   2. Discontinuation of other systemic SLE therapies (including mycophenolate and/or voclosporin)

   Exclusion Criteria for Cohort Extrarenal SLE:
10. Severe kidney disease as assessed locally, defined as history of ISN/RPS Class III to IV on renal biopsy.
11. Contraindication to methylprednisolone 500 mg daily for 2 days.
12. Any inability to discontinue or taper systemic SLE therapy prior to infusion of ATA3219, including

    1. Tapering of corticosteroids to ≤ 20 mg/day by Day -2, and
    2. Suspension of other systemic SLE therapies (including mycophenolate and/or voclosporin)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04-16 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-04-16 (Actual)

PRIMARY OUTCOMES:
Number of Participants With treatment-emergent adverse events, including adverse events of special interest | From administration of pretreatments (LD or methylprednisolone) through 90 days after administration of study drug
Number of Participants With Dose-limiting Toxicities | Day 1 through Day 28 of first dose of study drug
Maximum Tolerated dose | Day 1 through Day 28 of first dose of study drug
Recommended Phase 2 dose of ATA3219 | Day 1 through Day 28 of first dose of study drug

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of ATA3219 | Pre-dose on Day 1 through 24 months after the last dose on a defined schedule
Time to Reach Cmax (Tmax) of ATA3219 | Pre-dose on Day 1 through 24 months after the last dose on a defined schedule
Partial Area Under the Curve (pAUC) of ATA3219 | Pre-dose on Day 1 through 24 months after the last dose on a defined schedule
Last Observed Plasma Concentration (Clast) of ATA3219 | Pre-dose on Day 1 through 24 months after the last dose on a defined schedule
Time of Clast of ATA3219 | Pre-dose on Day 1 through 24 months after the last dose on a defined schedule
Terminal Half-life (t1/2) of ATA3219 | Pre-dose on Day 1 through 24 months after the last dose on a defined schedule
Complete Renal Response | Weeks 24 and 52
Partial Renal Response | Weeks 24 and 52
Renal Objective Response Rate | Weeks 24 and 52
Change From Baseline in Urine protein-to-Creatinine Ratio | Baseline (Day -5) through 24 months after the last dose on a defined schedule
Change From Baseline in Estimated Glomerular Filtration Rate | Baseline (Day -5) through 24 months after the last dose on a defined schedule
Duration of Urine Protein-to-Creatinine ratio ≤ 0.5 | Baseline (Day -5) through 24 months after the last dose on a defined schedule
Change From Baseline in Lupus Low Disease Activity State (LLDAS) | Baseline (Day 28) through 24 months after the last dose on a defined schedule
Change From Baseline in Definition of Remission in Systemic Lupus Nephritis (DORIS) | Baseline (Day 28) through 24 months after the last dose on a defined schedule
Change From Baseline in the Modified Version of the Safety of Estrogens in Lupus Erythematosus National Assessment version of the Systemic Lupus Nephritis Disease Activity (Hybrid SELENA-SLEDAI) Index | Baseline (Day 28) through 24 months after the last dose on a defined schedule
Change From Baseline in British Isles Lupus Assessment Group (BILAG) Index | Baseline (Day 28) through 24 months after the last dose on a defined schedule
Change From Baseline in SLE Responder Index (SRI)-4 | Baseline (Day 28) through 24 months after the last dose on a defined schedule
Change From Baseline in BILAG-based Composite Lupus Assessment (BICLA) Response | Baseline (Day 28) through 24 months after the last dose on a defined schedule
Change From Baseline in Antibodies to Double Stranded Deoxyribonucleic Acid | Baseline (Day -5) through 24 months after the last dose on a defined schedule
Change From Baseline in Complement Component 3 (C3) and Complement Component 4 (C4) Levels | Baseline (Day -5) through 24 months after the last dose on a defined schedule
Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) Activity Score | Baseline (Day 28) through 24 months after the last dose on a defined schedule
Number of Swollen and/or Tender Joints | Baseline (Day 28) through 24 months after the last dose on a defined schedule

CONTACTS AND LOCATIONS:
Overall Officials: Janal Urich, Study Director — Atara Biotherapeutics
Locations (1):
- Atara Biotherapeutics, Thousand Oaks, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petri M, Orbai AM, Alarcon GS, Gordon C, Merrill JT, Fortin PR, Bruce IN, Isenberg D, Wallace DJ, Nived O, Sturfelt G, Ramsey-Goldman R, Bae SC, Hanly JG, Sanchez-Guerrero J, Clarke A, Aranow C, Manzi S, Urowitz M, Gladman D, Kalunian K, Costner M, Werth VP, Zoma A, Bernatsky S, Ruiz-Irastorza G, Khamashta MA, Jacobsen S, Buyon JP, Maddison P, Dooley MA, van Vollenhoven RF, Ginzler E, Stoll T, Peschken C, Jorizzo JL, Callen JP, Lim SS, Fessler BJ, Inanc M, Kamen DL, Rahman A, Steinsson K, Franks AG Jr, Sigler L, Hameed S, Fang H, Pham N, Brey R, Weisman MH, McGwin G Jr, Magder LS. Derivation and validation of the Systemic Lupus International Collaborating Clinics classification criteria for systemic lupus erythematosus. Arthritis Rheum. 2012 Aug;64(8):2677-86. doi: 10.1002/art.34473. PMID 22553077
- [Background] Gordon C, Jayne D, Pusey C, Adu D, Amoura Z, Aringer M, Ballerin J, Cervera R, Calvo-Alen J, Chizzolini C, Dayer J, Doria A, Ferrario F, Floege J, Guillevin L, Haubitz M, Hiepe F, Houssiau F, Lesavre P, Lightstone L, Meroni P, Meyer O, Moulin B, O'Reilly K, Praga M, Schulze-Koops H, Sinico R, Smith K, Tincani A, Vasconcelos C, Hughes G. European consensus statement on the terminology used in the management of lupus glomerulonephritis. Lupus. 2009 Mar;18(3):257-63. doi: 10.1177/0961203308100481. PMID 19213865